CLINICAL TRIAL: NCT00611416
Title: The Role of Tea Catechins and Caffeine in Relation to Energy Metabolism in Man
Brief Title: The Role of Tea Catechins and Caffeine in Relation to Energy Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Unilever R&D (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: (KF) 01 279421; Unilever
Record Dates: First submitted 2007-08-21; First posted 2008-02-08 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Obesity
Keywords: catechins; caffeine; energy expenditure; fat oxidation; appetite
MeSH Terms: conditions — Obesity | interventions — Tea; Caffeine; epigallocatechin gallate; gallocatechol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Active treatment A
  Interventions: Dietary Supplement: green tea; Dietary Supplement: Mix of catechins and caffeine
- 2 (Experimental): Active treatment B
  Interventions: Dietary Supplement: green tea; Dietary Supplement: EGCG
- 3 (Experimental): Active treatment C
  Interventions: Dietary Supplement: green tea; Dietary Supplement: EGC
- 4 (Active Comparator): Positive control
  Interventions: Dietary Supplement: Caffeine
- 5 (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: green tea — different catechin combinations
  Arms: 1; 2; 3
Dietary Supplement: Mix of catechins and caffeine — 3 tablet a day
  Arms: 1
Dietary Supplement: EGCG — 3 tablets a day
  Other Names: epigallocatechin gallate
  Arms: 2
Dietary Supplement: EGC — 3 tablets a day
  Other Names: Epigallocatechin
  Arms: 3
Dietary Supplement: Caffeine — 3 tablets a day
  Arms: 4
Dietary Supplement: Placebo — 3 tablets a day
  Arms: 5

SUMMARY:
The aim of this study is to elucidate the role of specific catechins, a mixture of catechins and caffeine in relation to weight control with particular emphasis on energy metabolism and fat oxidation.

DETAILED DESCRIPTION:
Obesity is the result of an imbalance between energy intake (EI) and energy expenditure (EE). Thus, two ways to treat obesity are to reduce EI or increase EE. Bioactive food ingredients affecting energy metabolism, e.g. EE, fat oxidation, satiety and EI may help people to successfully control or manage their weight. Green tea, one of the most widely consumed beverages in the world, may possess beneficial effects on the treatment of obesity.

Green tea is made from the leaves of Camellia sinensis species of the Theaceae family. Green tea is the non- fermented/oxidised products, in contrast to black tea that is fully fermented/oxidised. Green teas contain high quantities of catechins and caffeine which are believed to be the active components affecting energy metabolism. EGCG is the most abundant catechin and has received the most attention (Yang et al., 2000). Caffeine represents approximately 3 to 5 % of the dry weight of green tea (Dufresne et al., 2001, Yang et al., 2000). It is general accepted that caffeine consumption is related to an increase in EE (Astrup et al., 1990), whereas the relation between catechins and energy metabolism is recently discovered.

In a study by Dulloo et al (1999), ten healthy men were assigned to 3 treatments: 1) green tea extract containing 150 mg/day caffeine and 270 mg/day of EGCG, 2) caffeine (150 mg/day) or 3) placebo. Ingestion of green tea extract (taken with each meal) increased 24-h EE by 4 % (328 kJ), reflecting its stimulatory effect on thermogenesis. This study also found a reduction in the respiratory quotient (RQ) during the green tea extract treatment, suggesting an increase in fat oxidation. However, Kovacs et al. (2004) did not report any changes in 24-h EE or RQ after same supplementation with green tea capsules, which may be explained by different background caffeine consumption.

Recently, two medium term studies have reported of increased fat oxidation after 8 and 12 weeks, respectively, supplementation with tea catechin containing beverage (Ota et al., 2005, Harada et al., 2005). In addition, Nagao et al. (2005) have shown that a daily consumption of tea beverage containing 690 mg/day catechins for 12 weeks reduced body fat area by 8% compared to the control group. Thus, catechins may not only promote EE, but also mildly reduce body fat.

Several potential mechanisms responsible for the altered energy and fat metabolism have been proposed. Dulloo et al. (1999) have suggested a synergistic interaction between catechins and caffeine due to sympathetically released noradrenaline (NA). Since catechins are known to be capable of inhibiting catechol O-methyltransferase (COMT) (the enzyme that degrades NA) (Borchardt & Huber, 1975), and caffeine to inhibit trancellular phosphodiesterases (enzymes that break down NA-induced cAMP), it is proposed that the green tea extract, via its catechins polyphenols and caffeine, is effective in stimulating thermogenesis by relieving inhibition at different control points along the NA-cAMP axis. Taken together, both caffeine and tea catechins would be expected to increase and/or prolong the stimulatory effects of norepinephrine on energy and lipid metabolism.

Several animal studies have been conducted to elucidate the anti-obese mechanisms of green tea extracts.

* Increased hepatic β-oxidation of fatty acids in mice after 4 weeks high fat diet with supplementation with tea catechins (74% EGCg, 18% ECg, 6% GCg, 2% others) (Murase et al., 2002 and 4 weeks high fat diet with supplementation with EGCg (Klaus et al., 2005). On the other hand, fatty acid synthase (FAS) was not altered by tea catechins, which may indicate that the simulation of fatty acid oxidation, rather than suppression of lipogenesis, is the predominant contribution (Murase et al., 2002).
* Modulated appetite and reduces food intake through the leptin receptor-independent pathway (Kao et al., 2000)
* Intraperitoneal administration of EGCg may reduce the diet digestibility resulting in increased faecal excretion of lipids (Klaus et al., 2005)
* Green tea extract (8% caffeine and 25% catechins (~70% EGCg)) stimulates brown adipose tissue thermogenesis and energy expenditure, which may be due to the prolonged effect of noradrenalin (Dulloo et al., 2000).

Large variations in catechin content and chemical structures occur during preparation and manufacturing of green tea products and therefore also among the studies. EGCg is the most intensely studied catechin. However, the plasma bioavailability of EGCg is lower than of EGC and EG (Henning et al., 2004), suggesting that non-galloylated catechins are better absorbed than the galloylated (Manach et al., 2005).

In addition, it is not known whether epimerization of catechins alters the effect on energy and fat metabolism (Harada et al., 2005, Ota et al., 2005, Xu et al., 2004). Therefore, it is not clear whether the reported effects are due to the total quantity of catechins, the chemical structure of specific catechins (e.g. epimerization and galloylation), and/or the caffeine content or other components of in the mix.

Methods

The study is a 5-way crossover double blind placebo controlled design. At each test day, energy expenditure and fat oxidation are measured via indirect calorimetry for 13 hours in one of two whole body respiratory chambers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* Age 18-40 years
* BMI 18,5-25 kg/m2

Exclusion Criteria:

* Diabetes or any other endocrinological disease
* Hypertensive medication
* Increased Blood Pressure > 140/85
* Hyperlpidimia
* Chronic disease (i.e. HIV)
* Use of any diet supplements including vitamins (during and 3 months prior to the study).
* High alcohol intake (>21 units a week)
* High caffeine intake (>250 mg/day) or high catechin intake (>200 mg/day)
* Smoking
* Elite sports performer
* Use of any regular medication

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
fat oxidation | november 2007

SECONDARY OUTCOMES:
appetite | november 2007

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Proffessor, Study Chair — Insitute of Human Nutrition
Locations (1):
- Institute of Human Nutrition, The Royal Veterinary and Agricultrual University, Frederiksberg C, Denmark